CLINICAL TRIAL: NCT05338944
Title: Dialectal Behaviour Therapy to Enhance Health Behaviour Change for Adolescents Living With Obesity (DIRECTION Trial)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Diabetes Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jon McGavock, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS24295
Record Dates: First submitted 2022-04-06; First posted 2022-04-21 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Prevention; Type2Diabetes

STUDY DESIGN:
Intervention Model Description: 90 youth will be randomized (2:2:1) into one of the three arms of the trial; DBT + lifestyle, lifestyle alone, control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- DBT + lifestyle (Experimental): Participants will receive 90 minutes of dialectical behavioral therapy and 90 minutes of lifestyle sessions each week for 16 weeks.
  Interventions: Behavioral: Dialectical behavioral therapy; Behavioral: Lifestyle
- Lifestyle alone (Experimental): Participants will receive 2 lifestyle sessions per week, 90 minutes each for 16 weeks.
  Interventions: Behavioral: Lifestyle
- Control (No Intervention): Participants will be included in baseline, endpoint and follow up measurements, but will receive no form of intervention.

INTERVENTIONS:
Behavioral: Dialectical behavioral therapy — Working with psychologists through DBT skills training.
  Arms: DBT + lifestyle
Behavioral: Lifestyle — Working with kinesiologist and registered dietician to improve lifestyle habits.
  Arms: DBT + lifestyle; Lifestyle alone

SUMMARY:
This research is being conducted to evaluate emotion-focused therapy that incorporates elements of mindfulness, distress tolerance, and relationship support. The investigators want to learn if this therapy, called Dialectical Behavioral Therapy (DBT) will help improve quality of life and weight management in youth at risk for type 2 diabetes. Individuals will be randomly assigned to weekly group based session in one of 3 intervention arms; lifestyle + DBT, lifestyle alone, or a control arm.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years old
* BMI z-score >1.4
* signs of mild-moderate depression (PHQ-9 score 5-19)
* willing and able to comply with study procedures

Exclusion Criteria:

* more than one health co-morbidity
* being treated with medication for obesity
* taking steroids
* currently being treated for atypical antipsychotics
* have an orthopedic injury or chronic illness that would prevent them from performing the intervention
* experienced weight loss or enrolled in weight loss program in the six months prior to the study
* they are currently and/or in the past 12 months have been prescribed any weight loss medication(s) including Ozempic
* self reported history of alcoholism or drug abuse
* history of self-harm or suicide attempts in the past 12 months
* currently enrolled in psychotherapy or DBT
* parents do not approve of you participating
* unable to read, speak and understand English as translation will not be provided
* unable/unwilling to give assent/consent

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-01-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Enrollment rates | 16 weeks
  defined as the number of adolescents/families who consent to participate and are randomized to one of the arms of the study
Adherence to the intervention | 16 weeks
  defined as the percentage of prescribed sessions that adolescents/families attend during the trial
Retention for follow up measurements | Measured at week 16 and week 32
  defined as the number of adolescents who complete follow up measurements at 16 weeks and 32 weeks

SECONDARY OUTCOMES:
Quality of Life measure using the PedsQL questionnaire | Measured at baseline, 16 weeks and 32 weeks
  Measure using the PedsQL questionnaire, subscales of emotional, social and health-related QOL will be treated separately and as a composite measure
Body composition measured by dual-x-ray absorptiometry (DXA) | Measured at baseline, 16 weeks and 32 weeks
  Measurements of % body fat, total fat, trunk fat, muscle mass, estimated VAT mass, estimated VAT volume and estimated VAT area will be collected, along with height and weight.
Body Mass Index (BMI) z-score | Measured at baseline, 16 weeks and 32 weeks
  Calculated using measured height and weight
Emotional regulation | Measured at baseline, 16 weeks and 32 weeks
  Measurement using the Difficulties in Emotion Regulation Scale (DERS) questionnaire.
Emotional reactive eating | Measured at baseline, 16 weeks and 32 weeks
  Measurement using the Child version of the Three-Factor Eating Questionnaire (TFEQ-R20 C).
Depressive symptoms | Measured at baseline, 16 weeks and 32 weeks
  Measured using the Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms.
Psychological distress | Measured at baseline, 16 weeks and 32 weeks
  Measured using the Kessler Emotional Distress Scale (K6) to assess psychological distress using six items covering depression and anxiety in the most recent 30 days.
Anxiety symptoms | Measured at baseline, 16 weeks and 32 weeks
  The parent and child version of the Screen for Child Anxiety Related Disorders (SCARED) questionnaire will be used to measure anxiety symptoms.
Readiness for Lifestyle Behavior Change | Measured at baseline, 16 weeks and 32 weeks
  Measured using the PACE readiness questionnaire which assesses readiness for changing dietary habits, daily activity goals and screen time.
Behavior regulation in exercise | Measured at baseline, 16 weeks and 32 weeks
  The BREQ3 (Behavioral Regulation in ExerciseQuestionnaire-3), will be used to measure of the level of motivation to engage in exercise from a self determination perspective.
Self-reported healthy lifestyle behaviors - physical activity and screen time | Measured at baseline, 16 weeks and 32 weeks
  Measured using the CANPWR questionnaire on physical activity and screen time habits.
  McPhee PG, Zenlea I, Hamilton JK, Ho J, Ball GDC, Mian R, Buchholz A, Laberge AM, Legault L, Tremblay MS, Chanoine JP, Thabane L, Morrison KM. Individual and family characteristics associated with health indicators at entry into multidisciplinary pediatric weight management: findings from the CANadian Pediatric Weight management Registry (CANPWR). Int J Obes (Lond). 2022 Jan;46(1):85-94. doi: 10.1038/s41366-021-00959-3. Epub 2021 Sep 9. PMID: 34504287.
Sleep habits | Measured at baseline, 16 weeks and 32 weeks
  The Sleep Disturbance Assessment Form (PROMIS) will be used to capture sleep habits.
Objective physical activity and sleep patterns | Measured at baseline, 16 weeks and 32 weeks
  A wrist worn fitbit will collect physical activity data and sleep data for 7 days at each timepoint. Data collected includes: steps per day, minutes of activity in low, moderate and high intensity, and total minutes of sleep per night.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Undecided